CLINICAL TRIAL: NCT02067364
Title: CRT ShuntCheck "Fit & Function" Exploratory Study
Brief Title: CRT ShuntCheck "Fit & Function" Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuroDx Development (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NDxDev-CRT-2015; R44NS074486 (NIH)
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Hydrocephalus
Keywords: hydrocephalus; CSF shunt
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fit & function test (Other): CRT ShuntCheck sensors will be applied over the shunts of asymptomatic hydrocephalus patients. The device will be activated, cooling the skin under the sensor. Patients will change positions during the one hour procedure and data will be recorded. Data will be analyzed offline to identify product performance issues due to motion.
  Interventions: Device: Fit & Function test

INTERVENTIONS:
Device: Fit & Function test
  Other Names: ShuntCheck; CRT ShuntCheck; ShuntCheck XM Extended Shunt Flow Monitor

SUMMARY:
An exploratory "Fit & Function" study of Continuous Real Time (CRT) ShuntCheck, a non-invasive method for monitoring changes in cerebrospinal fluid (CSF) shunt flow in hydrocephalus patients. The device will be tested on 10 pediatric patients (at Johns Hopkins Hospital) and 10 adult patients (at LifeBridge Health) and results will be used to optimize device design.

DETAILED DESCRIPTION:
An exploratory "Fit & Function" study of Continuous Real Time (CRT) ShuntCheck, a non-invasive method for monitoring changes in CSF shunt flow in hydrocephalus patients. This study will gather information to refine the design of the CRT ShuntCheck sensor. Our Aim I product work will yield a clinic-ready prototype which adheres well to human skin, conforms to the curve surface of the clavicle and provides a safe level of skin cooling over an extended period of time. Many of the clinical uses of CRT will involve patient movement - standing up to investigate suspected overdrainage, or the simple fidgeting of children undergoing monitoring. The Aim II Fit and Function testing will most importantly identify movement-related product performance issues. If we can identify the causes of "signal noise", we can modify our sensor design to make it less susceptible to "motion artifacts".

Additionally testing will identify age/size specific issues - is the sensor small enough for use on younger children, does the looser skin of older adults generate move motion artifacts in the signal.

These studies will include 10 pediatric and 10 adult asymptomatic patients who are willing to undergo CRT ShuntCheck testing over a one hour period. Test results will not be used to guide patient care and testing will not interfere with or delay any other patient testing or care.

ELIGIBILITY:
Inclusion Criteria:

1. For the pediatric subjects, males or females, older than three and less than 20 years of age.
2. For the adult subjects, males or females, older than 35 years of age
3. Parent/guardian or alert subject (age 18 or over) capable of giving consent; subject less than 18 and of assent age must give assent to participate if appropriate and required by the institution. If the subjects are incapable of giving assent, then only parent/guardian consent is required.
4. Possess an unambiguously identifiable chronically indwelling ventricular shunt which crosses the clavicle.

Exclusion Criteria:

1. Inability or unwillingness of the parent/guardian or alert subject to give informed consent/assent (when appropriate) as required by the Institutional Review Board.
2. Study testing would interfere with emergent subject care or if the subject is scheduled to go the OR in short order.
3. Presence of an interfering open wound or edema over the shunt.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Sensor fit & function | Single visit one hour test procedure
  Fit and Function testing will quantify the level and the duration of thermal changes due to patient movement compared with the level and duration of thermal changes due to changes in shunt flow. If motion related changes are > 0.5 times the level of flow related changes, the sensor and/or the procedure will be modified to improve signal to noise to >2.0

SECONDARY OUTCOMES:
Identify any safety issues | Single visit one hour test
  The CRT ShuntCheck test is a non-invasive, non-significant risk procedure. A small area of skin at the clavicle is cooled to and held at room temperature for an extended period of time. Study subjects should experience zero significant adverse events and no temperature related adverse events beyond minor discomfort. Any EA's will be addressed in design modifications.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - LifeBridge Health, Sinai Hospital of Baltimore (Testing Adult Patients 35 years+), Baltimore, Maryland
  - Johns Hopkins Hospital (Testing Pediatric Patients Age 3 to 19), Baltimore, Maryland